CLINICAL TRIAL: NCT01270113
Title: Improving Methadone Maintenance Treatment Compliance and Outcomes in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Yih-Ing Hser, Ph.D., Professor, Principal Investigator, UCLA Integrated Substance Abuse Programs
Other Study IDs: DESPR DA025252; 5R21DA025252-02 (NIH)
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2010-12

CONDITIONS: Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: contingency management

SUMMARY:
China faces the challenge of dual epidemics of drug use and HIV/AIDS. In responding to concerns of high rates of HIV/AIDS and other medical consequences among heroin users, China has recently implemented methadone maintenance treatment (MMT) programs nationwide. One problem noted with this rapid expansion is that the dropout rates from MMT have been high. The proposed study will adapt a motivational incentives (MI) intervention developed in the United States for use in Chinese MMT settings and will pilot test its effectiveness in improving treatment compliance and outcomes. The study's primary aims are: 1. to adapt a motivational incentives intervention in MMT in China, and 2. to experimentally pilot test the motivational incentives intervention. A secondary aim is to explore factors that may influence the outcomes of MMT that incorporates a motivational incentives intervention. It is hypothesized that the MI intervention can be adapted to Chinese settings and that it will optimize the positive outcomes of MMT in reducing HIV risks among heroin abusers. The collaborative team includes researchers in American and Chinese institutes (UCLA/Johns Hopkins/Washington, Shanghai Mental Health Center, Yunnan Institute for Drug Abuse), officials from national and local Chinese Centers for Disease Control and Prevention, and providers in local MMT clinics in Shanghai and Yunnan.

ELIGIBILITY:
Inclusion Criteria:adult patients entering the participating MMT clinics during the recruitment period who are dependent on heroin and who are willing to participate in the study.

Exclusion Criteria:Patients who are diagnosed with severe mental illness will not be eligible to participate.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult